CLINICAL TRIAL: NCT00006123
Title: Autotransplantation and Her 2 Neu Antibody Immunotherapy in Advanced Breast Cancer
Brief Title: Chemotherapy and Peripheral Stem Cell Transplantation Followed by Trastuzumab in Treating Women With Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Never started
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, David Avigan, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Purpose: Treatment
Other Study IDs: CDR0000068138; BIH-99-12; BIH-W-99-0053-FB; NCI-V00-1610
Record Dates: First submitted 2000-08-03; First posted 2004-02-12 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Carboplatin; Carmustine; Cisplatin; Cyclophosphamide; Thiotepa; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: trastuzumab
Drug: carboplatin
Drug: carmustine
Drug: cisplatin
Drug: cyclophosphamide
Drug: thiotepa
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Chemotherapy uses different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I/II trial to study the effectiveness of chemotherapy and peripheral stem cell transplantation followed by trastuzumab in treating women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and toxicity profile, specifically cardiac toxicity, of trastuzumab (Herceptin) following high dose chemotherapy and autologous peripheral blood stem cell transplantation in women with metastatic breast cancer. II. Determine the time to disease progression and disease free survival in these patients when treated with this regimen. III. Determine the impact of trastuzumab (Herceptin) on minimal residual disease after autologous peripheral blood stem cell transplantation as evidenced by serial immunocytochemical analysis of bone marrow. IV. Determine the relationship between posttransplant reconstitution of antibody dependent cellular toxicity and the efficacy of trastuzumab (Herceptin) in these patients.

OUTLINE: This is a multicenter study. Patients undergo stem cell mobilization with growth factors alone (filgrastim (G-CSF) and/or sargramostim (GM-CSF)) or chemotherapy followed by growth factors (depending on center). Peripheral blood stem cells (PBSC) are then collected by leukapheresis. Patients then receive high dose chemotherapy consisting of cyclophosphamide IV over 1 hour and cisplatin IV over 72 hours on days -6 to -4 and carmustine IV on day -3 or cyclophosphamide IV, thiotepa IV, and carboplatin IV over 96 hours on days -7 to -4 (depending on center). PBSC are reinfused on day 0. Patients then receive trastuzumab IV over 30-90 minutes weekly for 1 year or until disease progression beginning 5-8 weeks after PBSC reinfusion.

PROJECTED ACCRUAL: A total of 70 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage IV breast cancer that overexpresses HER2/neu Evidence of at least a partial response (at least 50% reduction) to salvage chemotherapy as initial chemotherapy for metastatic disease Measurable disease not required if there is no disease progression at induction chemotherapy Bone lesions as only site of metastatic disease allowed if evidence of clinical improvement and no new lesions on x-ray No CNS metastases Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 to physiologic 65 Sex: Female Menopausal status: Pre or postmenopausal Performance status: Karnofsky 80-100% Life expectancy: At least 6 months Hematopoietic: WBC at least 2,500/mm3 Absolute neutrophil count at least 1,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 2.5 times ULN Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: LVEF at least 45% by radionucleotide ventriculogram No uncontrolled hypertension No unstable angina No New York Heart Association class IV heart disease or congestive heart failure No coronary angioplasty or myocardial infarction within past 6 months No uncontrolled atrial or ventricular cardiac arrhythmias Pulmonary: FEV1 and DLCO at least 50% Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception HIV negative No insulin dependent diabetes mellitus No uncontrolled active systemic infection No other significant nonmalignant disease No other malignancy in past 5 years except surgically cured nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior trastuzumab allowed No prior bone marrow or peripheral blood stem cell transplantation Chemotherapy: See Disease Characteristics Prior doxorubicin not to exceed total cumulative dose of 360 mg/m2 No more than 6 standard courses of pretransplant salvage chemotherapy No more than 3 months of prior weekly taxane therapy More than 1 chemotherapy regimen allowed with no progression during chemotherapy Endocrine therapy: Concurrent tamoxifen therapy allowed for estrogen receptor positive patients who have not received prior hormonal therapy No other concurrent hormonal therapy Radiotherapy: No concurrent radiotherapy Surgery: Not specified Other: Concurrent pamidronate allowed for bone lesions

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2000-07; Primary Completion 2000-07 (Actual); Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Avigan, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey